CLINICAL TRIAL: NCT01846052
Title: Clinical and Genetic Characterization of Individuals With Achromatopsia
Status: Completed | Type: Observational
Sponsor: Beacon Therapeutics (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACHM-001; 1R24EY022023 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Achromatopsia
Keywords: achromatopsia, CNGB3
MeSH Terms: conditions — Color Vision Defects; Achromatopsia 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples will be stored at the DNA testing laboratory for additional testing for mutations in other genes that may be causally related to achromatopsia.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify individuals with achromatopsia caused by mutations in the CNGB3 gene and characterize their clinical condition using several tests of visual function every 6 months for up to 1.5 years.

DETAILED DESCRIPTION:
Individuals with a clinical diagnosis of achromatopsia will be asked to provide informed consent and will then have a single 5 mL blood sample drawn for DNA sequence analysis of genes known to cause achromatopsia, including the CNGB3 gene. All participants will be informed of the results of testing for these mutations. Those with mutations in both alleles of the CNGB3 gene will be evaluated every 6 months for up to 1.5 years by using a variety of non-invasive visual function tests to more fully characterize their clinical condition. This testing will include routine ophthalmic examination and tests of visual acuity, color vision, reading speed, perimetry, nystagmus, light sensitivity, optical coherence tomography, adaptive optics retinal imaging, electroretinography, fundus photography and completion of a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of achromatopsia (screening portion of study);
2. Molecular confirmation of mutations in the CNGB3 gene (main portion of study);
3. At least 6 years of age;
4. Willing and able to perform study procedures;
5. Signed informed consent(s) obtained (and child assent where applicable).

Exclusion Criteria:

1. Not able to have a blood sample drawn;
2. Pre-existing eye conditions that would interfere with interpretation of study endpoints (e.g. glaucoma, corneal or lenticular opacities, diabetic retinopathy, history of retinal detachment);
3. Participating in an interventional research study of drugs or devices for treatment of achromatopsia or other retinal diseases;
4. Use of medications that may impair color vision (e.g. hydroxychloroquine);
5. Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a clinical diagnosis of achromatopsia
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Annually for up to 1.5 years
  Visual acuity will be measured by EVA or ETDRS methods

SECONDARY OUTCOMES:
Color Vision | annually for up to 1.5 years
  Color vision will be measured by Farnsworth D-15 test and anomaloscope
Adaptive Optics Retinal Imaging | annually for up to 1.5 years
  Adaptive optics retinal imaging will be performed using the method of Genead et al. (Invest Ophthalmol Vis Sci 2011;52:7298-308).

CONTACTS AND LOCATIONS:
Overall Officials: Matt Feinsod, MD, Study Director — Applied Genetics Technologies Corporation
Locations (5):
- United States (5):
  - VitreoRetinal Associates, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Pangere Center for Inherited Retinal Diseases, The Chicago Lighthouse for People Who Are Blind or Visually Imp, Chicago, Illinois
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Langlo CS, Patterson EJ, Higgins BP, Summerfelt P, Razeen MM, Erker LR, Parker M, Collison FT, Fishman GA, Kay CN, Zhang J, Weleber RG, Yang P, Wilson DJ, Pennesi ME, Lam BL, Chiang J, Chulay JD, Dubra A, Hauswirth WW, Carroll J; ACHM-001 Study Group. Residual Foveal Cone Structure in CNGB3-Associated Achromatopsia. Invest Ophthalmol Vis Sci. 2016 Aug 1;57(10):3984-95. doi: 10.1167/iovs.16-19313. PMID 27479814